CLINICAL TRIAL: NCT02063711
Title: Acute Fetal Response to Prenatal Yoga: A Single Blinded, Randomized Controlled Trial (TRY Yoga Study)
Brief Title: Acute Fetal Response to Prenatal Yoga
Acronym: TRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Dev Maulik, MD, PhD, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13-941
Record Dates: First submitted 2014-01-30; First posted 2014-02-14 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Pregnancy
Keywords: Prenatal Yoga; Yoga, Pregnancy; Yoga, Fetal Response

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Intervention (Experimental): A 1-hour yoga session will take place with guided instruction provided by a registered yoga instructor. The class includes a warm up period of 5 minutes, which includes sitting with the eyes closed and slowly breathing through the nose. After which the participant will perform a series of yoga postures in coordination with her breathing for approximately 45 minutes. The last 10 minutes of class will encompass a semi-recumbent relaxation period. This is a one time intervention.
  Interventions: Behavioral: Yoga intervention
- Control group (No Intervention): In order to control for 1 hour worth of time, the participants in the control group will be given a 1 hour Power Point presentation on the benefits of exercise and yoga during pregnancy.

INTERVENTIONS:
Behavioral: Yoga intervention
  Arms: Yoga Intervention

SUMMARY:
Prenatal yoga has become a popular means of exercise during pregnancy.

DETAILED DESCRIPTION:
In 2012, yoga was reported to be practiced by approximately 20 million Americans, out of which 82% are women practitioners. The effects of yoga on the fetus have not been demonstrated. The purpose of this study is to evaluate the acute fetal response to yoga exercises by assessing fetal well-being via ultrasound and non-stress testing among healthy women. The investigators hypothesize that yoga during pregnancy does not have any acute negative effects on fetal behavior as assessed by umbilical artery Dopplers and fetal heart rate or maternal vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated singletons pregnancies
* Gestational age between 28 0/7 and 36 6/7 weeks
* No known fetal anomalies
* Women with no prior experience with yoga
* Currently receiving routine prenatal care
* No contraindications to exercise
* Able to read and understand English
* Well dated pregnancy

Exclusion Criteria:

* Pregnant minors less than 18 years of age
* Multiple gestations
* Those patients that have been advised by their doctor not to exercise during this pregnancy (i.e. Vaginal bleeding, history of preterm delivery less than 34 weeks, cervical insufficiency, cerclage in place, placenta previa, any chronic medical conditions)
* Congenital fetal anomalies or intrauterine growth restriction
* Cigarette smokers
* Chronic narcotic dependence

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
umbilical artery S/D ratio (Dopplers) | An umbilical artery ratio will be obtained on the day of intervention via an ultrasound machine. The first assessment will be before the intervention. The second assessment will be after a 1 hour intervention.
  The primary outcome of our study will be assessing umbilical artery S/D ratio (Dopplers). Doppler examination will be performed on the day of intervention. Approximately 20-30 minutes prior to the intervention and 20-30 minutes after a 1 hour intervention.

SECONDARY OUTCOMES:
Fetal Heart Rate | Fetal heart rate will be obtained on the day of intervention via a non stress test. The first assessment will be before the intervention. The second assessment will be after a 1 hour intervention.
  The secondary outcome will be the fetal heart rate. To assess if there is a change from 20-30 minutes prior to an intervention, to 20 -30 minutes after a 1 hour intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dev Maulik, MD, Principal Investigator — University of Missouri, Kansas City; Shilpa Babbar, MD, Study Director — University of Missouri, Kansas City
Locations (1):
- Truman Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Babbar S, Porter BW, Williams KB. The Impact of Prenatal Yoga on Exercise Attitudes and Behavior: Teachable moments from a Randomized Controlled Trial. Int J Yoga Therap. 2017 Nov;27(1):37-48. doi: 10.17761/1531-2054-27.1.37. PMID 29131740